CLINICAL TRIAL: NCT01736514
Title: A Randomized, Open Label, Multicenter, Allopurinol- Controlled Study to Assess the Safety and Efficacy of Oral Febuxostat in Patients With Gout
Brief Title: A Study to Evaluate Safety and Efficacy of Oral Febuxostat in Patients With Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMXALL-1001-TW
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Gout
Keywords: xanthine oxidase inhibitor; Uric acid lowering drug
MeSH Terms: conditions — Gout | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- febuxostat group (Experimental): oral
  Interventions: Drug: febuxostat
- allopurinol group (Active Comparator): oral
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: febuxostat — oral
  Other Names: Adenuric, Uloric, Feburic
  Arms: febuxostat group
Drug: Allopurinol — oral
  Arms: allopurinol group

SUMMARY:
This is a multicenter, open label, randomized, allopurinol-controlled, parallel-design study. Approximately 120 subjects will be randomly assigned in 1:1 ratio to receive febuxostat, or allopurinol for subjects with gout.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will also have a history or presence of gout as defined by the American College of Rheumatology (ACR) criteria
* Subject has serum urate level >= 8.0 mg/dL at the screening Visit

Exclusion Criteria:

* Female subject who is breast-feeding or pregnant
* Subject has a history of xanthinuria
* Subject who is intolerant of allopurinol, ie hypersensitivity, Steven-Johnson syndrome/topic epidermal necrolysis
* Subject who takes allopurinol > 300 mg/day and with serum urate level > 8mg/dL
* Subject who is HLA B*5801 positive
* Subject who is receiving thiazide diuretic therapy
* Subject who has secondary hyperuricemia
* Subject who requires concurrent therapy with any systemic or topical medications, prescribed or non-prescribed, containing aspirin or other salicylates (low doses of aspirin will be allowed(ie. =< 325mg/day)
* Subject who requires therapy with prednisone > 10 mg/ day during the study
* Subject who has active liver disease or hepatic dysfunction, defined as both ALT and AST > 1.5 times the upper limit of normal
* Subject who has serum creatinine >= 1.5mg/dL
* Subject who has any another significant medical condition as defined by the investigator that would interfere with the treatment, safety or compliance with the protocol (eg. A clinically significant ECG result)
* Subject who has a history of cancer (other than basal cell carcinoma of the skin) within 5 years prior to the study, or has taken any systemic cancer chemotherapy within 5 years prior to the study
* Subject who has previously participated in a clinical study in which febuxostat was administered
* Subject who has participated in another investigational trial within the 30 days prior to the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects whose serum urate level decreases to < 6.0 mg/dL | week 12

SECONDARY OUTCOMES:
Percent reduction in serum urate levels | Baseline and at week 12
Safety assessed by the incidence of adverse events, physical exam. and vital signs, tabo-tests and 12-lead ECG | Baseline and at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Taiwan, Inc.
Locations (4):
- Taiwan (4):
  - Kaohsiung City
  - Linkou District
  - Taichung
  - Taipei